CLINICAL TRIAL: NCT02512159
Title: Effectiveness of Topical Negative Handicraft Device for Versus Traditional Conservative Treatment in Skin Ulcers Management in Lower Limb
Brief Title: Skin Ulcers Treatment With an Handicraft Topical Device
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-2301-12
Record Dates: First submitted 2015-03-12; First posted 2015-07-30 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2014-02

CONDITIONS: Foot Ulcer; Varicose Ulcer
Keywords: Diabetic foot ulcer; Foot care; Wound management
MeSH Terms: conditions — Foot Ulcer; Varicose Ulcer; Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- drenovac handcrafted (Experimental): Patients treatment with the handicraft topical device negative pressure therapy Economic craft
  Interventions: Procedure: drenovac handcrafted
- Healing (Active Comparator): Patients who were managed with traditional "conservative treatment".
  Interventions: Procedure: Healing

INTERVENTIONS:
Procedure: drenovac handcrafted — under local anesthesia, sepsis and antisepsis, place sterile field, prepared area go out all devitalized or necrotic tissue using liquid soap surgical and irrigation back saline 0.9%. We introduce a device to distribute the negative pressure or vacuum on ulcer; conducted margins make recommendations 5-12 mm over the edge of the wound, applying negative pressure or vacuum retracted sponges, likewise for the spare fewer gauze was placed Sterile adhesive film covering the defect to seal the system cover adequately the probe output nelaton not to submit drain the system. Connect the probe to the sterile nelaton this hose and a suction system with pressure gauge, pressure -80-125 mmHg. Change it every 72 hours.
  Arms: drenovac handcrafted
Procedure: Healing — Were handled as follows:
  1. Under local anesthesia, prior asepsis and antisepsis of the skin ulcer with iodinepovidone sterile fields are placed, we proceeded to debridement of all necrotic tissue or devitalized then a cure with liquid soap surgery was performed and was irrigated with 1000 cc of solution physiological 0.9%, and finally the ulcer was covered with sterile gauze.
  2. healing of skin ulcers were performed every 24 hours.
  3. the evolution of skin ulcers was evaluated every 3 days, requesting a differential valuing of clinical and biochemical form the aforementioned variables.
  Arms: Healing

SUMMARY:
The aim of this study was to evaluate the efficacy of a handicraft topical device of negative pressure versus traditional healing treatment for skin ulcers in lower limbs; in patients with diabetes mellitus, venous stasis and arterial insufficiency.

DETAILED DESCRIPTION:
The hypothesis of this trial is that the handicraft topical device of negative pressure is even better for the treatment of skin ulcers located in the lower limbs of patients with diabetes mellitus, venous stasis and arterial insufficiency. We anticipate that in a sample of 144 patients with ulcer, will heal or at least improve with this treatment

ELIGIBILITY:
Inclusion Criteria:

1. Patients with cutaneous leg ulcers due to diabetes mellitus, venous stasis and arterial insufficiency requiring healing or tissue debrided sent to managing their disease to regional general hospital No. 17, Instituto Mexicano del Seguro Social, Benito Juárez, Quintana Roo.
2. Patients of both sexes.
3. Patients over 18 years.
4. Patients that have basic laboratory at admission (complete blood count with differential).
5. Patients with comorbidities associated as Diabetes Mellitus , Hypertension, stroke, heart disease, nephropathy, venous insufficiency and arterial insufficiency, etc.

Exclusion Criteria:

1. Hemodynamically unstable patients.
2. Patients with septic shock from any source.
3. Patients with deep skin ulcers with exposed some organ, data osteomyelitis, vascular-nervous exposure.
4. Patients with secondary cutaneous ulcer enteral fistula.
5. Patients with cutaneous ulcer or cancer tumors.
6. Patients with cutaneous ulcer with active bleeding.
7. Patients with cutaneous ulcer necrosis.
8. Patients with cutaneous ulcer leishmania, insect bite.
9. Patients with cutaneous ulcer burns.
10. Patients who do not accept their participation in the study through informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Presence of granulation tissue in skin ulcers. | 10 days
  Presence of granulation tissue in 50% of the wound

SECONDARY OUTCOMES:
Leukocyte less than 11,000 mm3. | 10 days
  Leukocyte less than 11,000 mm3.
Temperature | 10 days
  less than 38 ° C temperature.
Breathing Rate | 10 days
  less than 20 rpm breathing rate.
Heart Rate | 10 days
  lower heart rate 90 bpm.

CONTACTS AND LOCATIONS:
Overall Officials: Fany Guadalupe Pat Espadas, MCs, Principal Investigator — IMSS; Israel Augusto González González, Dr., Study Chair — IMSS; Luis Sandoval Jurado, PhD, Study Director — IMSS; Ma. Valeria Jiménez Baéz, PhD, Study Chair — IMSS

REFERENCES:
- [Derived] Gonzalez IG, Angel MA, Baez MV, Ruiz Flores B, de Los Angeles Martinez Ferretiz M, Woolf SV, Lopez I, Sandoval-Jurado L, Pat-Espadas FG, Cruz AA, Delgado AT. Handcrafted Vacuum-Assisted Device for Skin Ulcers Treatment Versus Traditional Therapy, Randomized Controlled Trial. World J Surg. 2017 Feb;41(2):386-393. doi: 10.1007/s00268-016-3782-9. PMID 27822727